CLINICAL TRIAL: NCT00585975
Title: Efficacy and Safety of Bromfenac Ophthalmic Solution
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CL-S&E-0802071-P
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Results first posted 2011-12-09 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Cataract Surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bromfenac Ophthalmic Solution 0.18% (Experimental)
  Interventions: Drug: bromfenac ophthalmic solution
- Xibrom 0.09% (Experimental)
  Interventions: Drug: bromfenac ophthalmic solution

INTERVENTIONS:
Drug: bromfenac ophthalmic solution — sterile opthalmic solution

SUMMARY:
This is a safety and efficacy study of bromfenac ophthalmic solution

ELIGIBILITY:
Inclusion Criteria:

* Male or female greater than or equal to 18 years of age, and scheduled for cataract surgery

Exclusion Criteria:

* Active corneal pathology in either eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim McNamara, PharmD, Study Director — ISTA Pharmaceuticals, Inc.
Locations (1):
- ISTA Pharmaceuticals, Inc., Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bromfenac Ophthalmic Solution 0.18% | Xibrom 0.09%
Started | 277 | 291
Completed | 262 | 278
Not Completed | 15 | 13
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Lost to Follow-up | 2 | 1
Not completed — Enrollment met/over-enrolled | 10 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bromfenac Ophthalmic Solution 0.18% | Xibrom 0.09% | Total
Number analyzed (Participants) | 277 | 291 | 568
Age Continuous [Mean (Full Range); unit: years] | 68.8 [37 to 90] | 68.6 [41 to 90] | 68.7 [37 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169 | 154 | 323
  Male | 108 | 137 | 245

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Summed Ocular Inflammation Score (SOIS) of Zero
Description: Participants with SOIS of 1. Scale: 0=0 cells (complete absence); 0.5=1-5 cells (trace); 1=6-15 cells (very slight); 2=16-25 cells (moderate); 3=26-50 cells (marked); 4=>50 cells (intense)
Time Frame: Day 15
Measure: Number; unit: Participant
Arm/Group | Bromfenac Ophthalmic Solution 0.18% | Xibrom 0.09%
Number analyzed (Participants) | 277 | 291
Participant | 157 | 164

2. Secondary Outcome: Number of Participants That Are Pain Free
Description: Participant description of being pain free taken from patient questionnaire with multiple possible responses
Time Frame: Day 1
Measure: Number; unit: Participant
Arm/Group | Bromfenac Ophthalmic Solution 0.18% | Xibrom 0.09%
Number analyzed (Participants) | 277 | 291
Participant | 221 | 235

ADVERSE EVENTS:
Arm/Group | Bromfenac Ophthalmic Solution 0.18% | Xibrom 0.09%
Serious Adverse Events (participants affected / at risk) | 2/266 | 3/278
Other Adverse Events (participants affected / at risk) | 13/266 | 19/278
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bromfenac Ophthalmic Solution 0.18% (N=266) | Xibrom 0.09% (N=278)
Skin Necrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Abnormal Skin Odor (Skin and subcutaneous tissue disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Anterior Chamber Inflammation (Eye disorders) | 0 | 1
Upper Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Kidney Infection (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bromfenac Ophthalmic Solution 0.18% (N=266) | Xibrom 0.09% (N=278)
Conjunctival Hyperaemia (Eye disorders) | 13 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI will provide to the sponsor a copy of the proposed publication information for review, comment and approval following completion of the study and at least sixty (60) days prior to submission for publication of any manuscript, or at least thirty (30) days prior to submission for publication of any abstract. If sponsor requests in writing, the PI will withhold publication for an additional sixty (60) days.